CLINICAL TRIAL: NCT05177991
Title: The Evaluation of Post-operative Pain Control With a TAP Block Using Exparel vs. Marcaine for Hernia Repairs
Brief Title: Post-operative Pain Control-TAP Block Using Exparel vs. Marcaine for Hernia Repairs
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Leslie Son (Other)
Collaborators: Our Lady of the Lake Hospital (Other)
Responsible Party: Sponsor-Investigator, Leslie Son, Research Scientist, Our Lady of the Lake Hospital
Organization: Our Lady of the Lake Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Anesthesia_Hernia_Pain
Record Dates: First submitted 2021-12-02; First posted 2022-01-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Inguinal Hernia; Ventral Hernia
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Ventral | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Single Blind, randomized
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine (Exparel) (Active Comparator): The bilateral TAP block will be performed by the department of anesthesia under ultrasound guidance using 20cc of local anesthetic per side. Additional local anesthetic will be supplied by the surgeon at the incision sites.
  Interventions: Drug: Liposomal Bupivacaine
- Bupivacaine (Marcaine) (Active Comparator): The bilateral TAP block will be performed by the department of anesthesia under ultrasound guidance using 20cc of local anesthetic per side. Additional local anesthetic will be supplied by the surgeon at the incision sites.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Liposomal Bupivacaine — 20cc of Liposomal Bupivacaine for TAP block
  Arms: Liposomal Bupivacaine (Exparel)
Drug: Bupivacaine — 20cc of Bupivacaine for TAP block
  Arms: Bupivacaine (Marcaine)

SUMMARY:
While studies have shown improved postoperative pain control with TAP blocks after inguinal and ventral hernia repair, data comparing Liposomal bupivacaine (Exparel) to bupivacaine alone in formulation of the TAP block is particularly scarce. Therefore, we designed a prospective, randomized trial comparing the postoperative pain control in minimally invasive ventral and inguinal hernia repair patients who receive an Exaparel-based TAP block compared to the traditional bupivacaine (Marcaine) TAP block.

DETAILED DESCRIPTION:
Approximately 200 patients in the study will be randomized to one of two arms: TAP block with Exparel or TAP block with bupivacaine. Randomization will be performed using a permuted block randomization algorithm (Ex. AABBABABABBABBAA, where A=Exparel group and B=Bupivacaine group). Only the participant will be blinded to the arm assignment as the knowledge of the assignment for the surgeon and anesthesiologist is needed. The bilateral TAP block will be performed by the department of anesthesia under ultrasound guidance using 20cc of local anesthetic per side. Additional local anesthetic will be supplied by the surgeon at the incision sites. Both of these anesthetics being evaluated and the dosage are commonly administered as standard of care (SOC). The choice of anesthetic used is up to the discretion of the surgeon in most instances. The patients will be blinded to which local anesthetic they receive. Operative technique will be standardized amongst all participating surgeons.

All patients with ventral hernias will undergo an IPOM+ technique detailed by primary closure of the defect in addition to circumferential mesh fixation with a running suture. Three or four trochars will be used ranging from 5-12mm in size. Mesh selection will be at the discretion of the surgeon with a minimum of 5cm overlap of the original defect in all directions. Defect size will be measured intraoperatively with a ruler intra-abdominally.

All patients with an inguinal hernia will undergo a transabdominal preperitoneal hernia repair with mesh placement. Three or four trochars ranging from 5-12mm will be used. Size of mesh and fixation of mesh at one or two points will be at the surgeon's discretion. The length of surgery will be recorded.

The patients will be given a packet of VAS pain assessments to take home with pre-marked time intervals to fill out at 2h, 6h, and 12h post operatively as well as every 12 hours thereafter. The patients will also be asked to record how many narcotic medications they will be consuming on a daily basis. Our team will contact patients daily to collect the data verbally which will also serve as a reminder to patients to complete this task faithfully. Each patient will follow up at one week and provide the surgeons with the packet of VAS assessments as well as bring in any excess narcotics that they did not consume. Each patient will also be told to take tylenol 500mg every 6 hours for the first 96 hours and to record whether they take any additional alternative pain medications (NSAIDs, muscle relaxants, gabapentinoids). Upon discharge, patients will be prescribed 15 pills of 5mg hydrocodone-325mg acetaminophen to be taken every 6 hours as needed for severe pain.

Data collection will include demographics of the patients including age, sex, ASA status, height/weight, BMI, preoperative pain level and previous abdominal surgeries. Intraoperative variables will include defect size, ventral vs. inguinal, number of trochar, mesh size and type, operative time. Postoperative collection will include pain scores as outlined above and narcotic use. Data analysis will include differences, if any, in post operative pain scores as well as narcotic use. This will be stratified to the inguinal hernia group vs. ventral hernias and the ventral hernia group will be stratified to size of defect and length of surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have a ventral or inguinal hernia requiring surgical repair

Exclusion Criteria:

* Less than 18 years of age
* Chronic pain patients
* Having a defect >10 cm in transverse dimension
* Having a defect <4 cm
* Has an allergy to bupivacaine
* Has recurrent hernias as per medical history
* A TAP block performed at any time aside from just prior to the start of the procedure
* If bupivacaine is mixed with other anesthetics
* Under the instance of an emergency surgery (trauma)
* Concomitant surgery
* History of EtOH abuse
* History of liver/kidney dysfunction
* If the procedure must be converted to open
* Inidividual's weight < 50kg
* Individual's BMI > 45

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Pain Scores using Visual Analog Scale (VAS) | For 1 week post-operation
  Lower mean daily post-operative pain scores between participants in the Exparel vs. Bupivacaine arms recorded multiple times over the observation period. The pain scale is 0-10 with 0 being no pain to 10 being the worst pain possible.

SECONDARY OUTCOMES:
Opioids Used Post-Operatively compared in anesthesia arms | For 1 Week post-operation
  The amount of opioid pills taken, as measured by morphine equivalents, is reduced depending on the type of anesthetic used during the TAP block. We will be measuring the post operative opioid usage by asking the patients how many narcotic pills they take daily after surgery for one week. Variability comes into play if we prescribe different doses of Norco or if we use Percocet, therefore we will standardize this by converting these differing dosages in to morphine equivalents for both groups.
Opioids Used Post-Operatively related to Hernia Size and Surgical Time | After 1 week post-operation
  A decrease in the total number of opioid pills taken post-operatively compared to the total surgical time and how large the hernia defect is. Increased surgical times and larger hernias may play a role in the amount of pain medication an individual may need post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Son, PhD, Study Director — Our Lady of the Lake Hospital
Locations (1):
- Karl LeBlanc, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No